CLINICAL TRIAL: NCT02619786
Title: Therapy of Ventilator-associated Tracheobronchitis Caused by Gram Negative Bacteria With Nebulized Colistin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Adhiratha Boonyasiri, Dr., Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 512-2558-EC4
Record Dates: First submitted 2015-11-26; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Bronchitis
MeSH Terms: conditions — Bronchitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- inhaled colistin (Experimental): Inhaled colistin 75 mg mixed with normal saline up to 4 ml every 12 hours at least 5 days
  Interventions: Drug: Inhaled colistin

INTERVENTIONS:
Drug: Inhaled colistin — 75 mg of colistin activity, inhaled per dose, every 12 hours
  Other Names: Colistate 150

SUMMARY:
The purpose of this study is to determine whether inhaled colistin is effective in the treatment of ventilator associated tracheobronchitis due to gram negative organism susceptible to colistin.

DETAILED DESCRIPTION:
Patients diagnosed ventilator-associated tracheobronchitis due to gram negative organism are included to the study.The patients will be received colistin inhalation 75 mg every 12 hours at least 5 days.

The primary objective is to evaluate clinical outcome of inhaled colistin. The secondary objectives are microbiological clearance and toxicity of inhaled colistin.

The sample size was estimated to 62 patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ventilator-associated tracheobronchitis caused by gram negative organism.
* Expected to survive more than 48 hours after enrollment.
* Received intravenous colistin not more than 48 hours prior enrollment.

Exclusion Criteria:

* Pregnancy and Lactation
* Allergy to colistin
* Serum creatinine > 4 mg/dl or GFR decreased more than 75% from baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of Patients With Cure, Improved, Failure or Death | through study completion, an average of 2 weeks
  Clinical outcome is classified in 4 categories:
  Cure Improved Failure Death

SECONDARY OUTCOMES:
Number of Patients With Eradication, Persistence or Superinfection | through study completion, an average of 2 weeks
  Microbiological response is classified in 4 categories:
  Eradication Persistence Superinfection
Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug, Graded According to NCI CTCAE Version 3.0 | through study completion, an average of 2 weeks
  Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug, Graded According to NCI CTCAE Version 3.0 focus on neurology and bronchospasm. Nephrotoxicity uses RIFLE criteria for acute kidney injury. RIFLE is an acronym of Risk, Injury, and Failure; and Loss; and End-stage kidney disease.

REFERENCES:
- [Background] Rattanaumpawan P, Lorsutthitham J, Ungprasert P, Angkasekwinai N, Thamlikitkul V. Randomized controlled trial of nebulized colistimethate sodium as adjunctive therapy of ventilator-associated pneumonia caused by Gram-negative bacteria. J Antimicrob Chemother. 2010 Dec;65(12):2645-9. doi: 10.1093/jac/dkq360. Epub 2010 Sep 28. PMID 20876621